CLINICAL TRIAL: NCT05598359
Title: TA-65 and Aging Associated Microvascular Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Louisville (Other); Penn State University (Other)
Responsible Party: Principal Investigator, William Hughes, Postdoc Fellow, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TA-65 and Vascular Aging
Record Dates: First submitted 2022-10-18; First posted 2022-10-28 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Telomere Shortening; Aging; Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TA-65 (Experimental): TA-65 (250 U) taken once per day
  Interventions: Dietary Supplement: TA-65
- Placebo (Placebo Comparator): Placebo taken once per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: TA-65 — TA-65 is a purified small molecule extracted from Astragalus root
  Arms: TA-65
Other: Placebo — Inactive formulation
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test whether activation of telomerase with a dietary supplement (TA-65) improves microvascular function.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to examine whether activation of autophagy with TA-65 which activates telomerase, improves microvascular function and blood pressure in an older population

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults 18 - 35 and 65+ years of age
* Subjects with clinical diagnosis of CAD

Exclusion criteria will include:

* 36-64 years of age without clinical diagnosis of CAD
* Self-reported habitual vigorous exercise (>20 min, 3 times per week, 1 yr)
* Major Adverse Cardiovascular Event (MACE) in the last year (heart attack, stroke)
* Heart Failure
* Renal Impairment
* >3 Pre-existing Cardiovascular Risk Factors (healthy groups only)
* Type 1 or type 2 diabetes
* Uncontrolled hypertension
* Current tobacco use or within last 6 months
* BMI > 35
* Hyperlipidemia
* Hypercholesterolemia
* Use of anti-coagulant drugs
* Use of anti-platelet drugs
* Erectile dysfunction medication in the past 6 months
* Use of topical/non-topical steroids in last 6 months
* Hormone replacement therapy (Post-Menopause or Gender Reassignment)
* History of retinopathy
* Documented neuromuscular disorders
* Porphyria Cutanea Tarda (blistering of skin to sun; photosensitivity)
* Pregnancy (young female subjects)
* Allergy to lidocaine
* Current diagnosis of cancer with or without active anti-cancer treatment (pharmaceuticals) or treatment within last 12 months
* Active COVID-19 or within the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Nitric Oxide Mediated Endothelium-Dependent Vasodilation via Laser Doppler Flowmetry Coupled with Intradermal Microdialysis | 28 days
  Cutaneous microvascular function measured via laser Doppler flowmetry coupled with intradermal microdialysis of non-specific nitric oxide synthase inhibitor, L-NAME

SECONDARY OUTCOMES:
Systemic Blood Pressure | 28 days
  Brachial systolic, and diastolic blood pressure will be measured via standard brachial blood pressure cuff

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Beyer, Ph.D., Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data available upon record completion